CLINICAL TRIAL: NCT04774978
Title: Real-time Automatic Continuous Cardiac Output Measurements Using Transthoracic Echocardiography (TTE) in ICU-patients in Comparison to Flotrac Measurements
Brief Title: Real-time Continuous Cardiac Output Measurements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RijnstateH
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Output, Low
Keywords: Cardiac output; TTE
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cardiac output measurements (Experimental): Cardiac output will be measured using TTE continuously with ProbeFix
  Interventions: Device: TTE

INTERVENTIONS:
Device: TTE — Transthoracic echocardiography

SUMMARY:
Study to assess the feasibility of real-time automatic cardiac output measurements using transthoracic echocardiography (TTE)

DETAILED DESCRIPTION:
Rationale: Study to assess the feasibility of real-time automatic cardiac output measurements using transthoracic echocardiography (TTE)

Objective: To assess the correlation and feasibility of real-time automatic continuous cardiac output measurements using transthoracic ultrasound (TTE) in adult ICU-patients in comparison to Flotrac measurements

Study design: prospective, feasibility study

Study population: Adult Intensive Care patients ( > 18 years)

Intervention (if applicable):

Consecutive adult patients on the ICU in which the there is an indication for continuous cardiac output measurements.

Main study parameters/endpoints:

* Percentage of patients in which continuous cardiac output can be measured using TTE
* Correlation between continuous TTE and Flotrac measurements

ELIGIBILITY:
Inclusion Criteria:

* Adult Intensive Care patients ( > 18 years)

Exclusion Criteria:

* Pregnancy
* Atrial fibrillation or other irregular heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Patients in which the ProbeFix can be used continuously | 2 months
  Percentages will be reported

SECONDARY OUTCOMES:
Correlation between continuous TTE and Flotrac | 2 months
  Bland-Altman plot will be reported